CLINICAL TRIAL: NCT04955366
Title: Late Abatacept Conversion in Kidney Transplant Recipients Receiving Belatacept: a Prospective, Randomized Controlled Non-inferiority Trial. IM101-884
Brief Title: Abatacept Conversion in Kidney Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Idelberto Badell, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001855
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Renal Transplant Recipient
Keywords: Renal transplant
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Belatacept group (Control Group) (Active Comparator): Participants will receive the following:
  * Belatacept: 5 mg/kg i.v. monthly
  * Blood draws for PD studies at baseline/Month 0 and Month 6 fora total of two timepoints.
  * HLA labs at 6, 12 and 24 months
  * Basic chemistry panel (CP Basic) every 3 months per clinical protocol for efficacy analysis
  * Hemoglobin A1c at Screening visit
  * Urine pregnancy test via test kit for WOCP at Screening visit
  * BK and CMV testing at 6, 12, and 24 months
  Interventions: Drug: Belatacept
- Abatacept Group (Conversion Group) (Experimental): Participants will receive the following:
  * Abatacept 125 mg s.c. weekly
  * Safety labs every 2 weeks (months 0-3) then monthly (months 4-12)
  * Blood draws forPK atMonth 6, Month 12, and two random time points in between Month 6 and Month 12 for a total of four time points.
  * Blood draws for PD studies at baseline/Month0 and Month 6 fora total of two timepoints.
  * HLA labs at 6, 12 and 24 months
  * Basic chemistry panel (CP Basic) at each study visit per clinical protocol for efficacy analysis
  * Hemoglobin A1c at Screening visit
  * Urine pregnancy test via test kit for WOCP at screening
  * BK and CMV testing at 6, 12, and 24 months
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Belatacept — Belatacept is an immunosuppressive medication and will be given as an intravenous infusion at a dose of 5 mg/kg monthly
  Other Names: Nulojix
  Arms: Belatacept group (Control Group)
Drug: Abatacept — Abatacept is an immunosuppressive medication and will be given SQ at a dose of 125 mg s.c. weekly
  Other Names: Orencia
  Arms: Abatacept Group (Conversion Group)

SUMMARY:
This is a single center, randomized, controlled phase 2b, conversion trial. This protocol has been developed to answer the question: Can patients be safely converted from monthly belatacept IV infusions to abatacept subcutaneous injections without a decrease in kidney function.The primary objective will be the difference in estimated GFR (eGFR) for abatacept and belatacept groups using a monthly repeated measures model between randomization and 12 months.

DETAILED DESCRIPTION:
This is a single center, randomized, controlled phase 2b, conversion trial. This protocol has been developed to answer the question: Can patients be safely converted from monthly belatacept IV infusions to abatacept subcutaneous injections without a decrease in kidney function. Research subjects will be recruited from those who were initiated on belatacept at the time of their kidney transplant and have been stable on belatacept therapy for at least 2 years post-transplant and off CNI therapy for at least 6 months.

A total of 86 subjects will be randomized in equal numbers, 43 patients in each arm. Enrollment of all 86 patients is expected to be completed within 1.5 years. All patients will be actively followed in the study for 24 months following randomization. The patient participation is projected to last a total of 3.5 years with data analysis to follow.

The primary objective will be the difference in estimated GFR (eGFR) for abatacept and belatacept groups using a monthly repeated measures model between randomization and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

1. Adult (age ≥18 years currently)
2. First-time renal transplant recipients of either living donor or deceased donor

   1. Treatment with belatacept from the time of transplant
   2. At least 2 years post-transplant and off CNI therapy for at least 6 months
3. Patients at low immunologic risk

   1. First time transplant
   2. HLA antibody screen with PRA < 80% against class I and class II antigens
   3. Negative crossmatch (actual or virtual)
   4. No donor specific anti-HLA antibody (DSA)
   5. No more than one episode of rejection (Banff grade 1A or greater)
   6. No episodes of rejection (borderline or greater) within the last 6 months prior to study participation
   7. No rejection of Banff grade IIB or greater
4. Immunosuppression consisting of belatacept (5mg/kg q 1M), mycophenolate mofetil (at least 1000 mg daily), or equivalent mycophenolic acid (720 mg daily) or azathioprine (1- 2 mg/kg daily) dose, and prednisone 5 mg daily.
5. Confirmed Tb screening at the time of transplantation

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

1. Repeat renal transplant, or multi-organ transplant recipient
2. History of more than one episode of biopsy-proven acute rejection (Banff grade 1A or greater), or of any episode of rejection of Banff 97 grade IIB or greater, or any rejection (borderline or greater) within the last 6 months
3. Pregnancy (women of childbearing potential must use adequate contraception during study)
4. GFR less than 35
5. Serum creatinine at enrollment more than 30% higher than at 3 months (±4 weeks) prior to randomization
6. Recent history of clinically significant proteinuria (urinary protein/Cr ratio >1.0)
7. Receiving belatacept at a dose other than 5 mg/kg body weight
8. Receiving mycophenolate mofetil at a dose of less than 1000 mg po QD (or mycophenolic acid or azathioprine equivalent).
9. Receiving prednisone at a dose greater than 5 mg po qd within 3 months of enrollment
10. Not currently receiving maintenance immunosuppression with prednisone
11. Active infection, or antibiotic or antiviral drug therapy within 1 month of randomization
12. Evidence of CMV viremia or clinical CMV infection within the last 3 months prior to randomization.
13. BK viremia of greater than 4.3 DNA log copies/mL (greater than 20,000 copies/mL) within 3 months of randomization
14. Known hepatitis B surface antigen-positive or PCR-positive for hepatitis B (testing not required)
15. Known HIV-positivity (testing not required)
16. Presence of donor specific antibody by Luminex single antigen bead assay, or antibody screen (% PRA) above 80%.
17. History of substance abuse or psychiatric disorder not compatible with study adherence and follow up.
18. History of medical noncompliance
19. Untreated latent Tb (as determined from prior Tb screening at the time of transplantation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in mean estimated GFR (eGFR) between randomization and 12 months post baseline | Baseline, 12 months post baseline
  Difference in estimated GFR (eGFR) for abatacept and belatacept groups using a monthly repeated measures model between randomization and 12 months.

SECONDARY OUTCOMES:
Change in eGFR between abatacept and belatacept groups at 24 months | Monthly until 24 months post baseline
  The treatment difference in eGFR between abatacept and belatacept groups at 24 months, using a monthly repeated measures model and a pre-specified acceptable difference, or non-inferiority margin of 5 ml/min/1.73m2.
Number of subjects with biopsy proven acute rejection: Acute Cellular Rejection (ACR) | 12 months post baseline, 24 months post baseline
  Incidence and severity of acute cellular rejection (ACR)
Number of subjects with biopsy proven acute rejection: Antibody Mediated Rejection (AMR) | 12 months post baseline, 24 months post baseline
  Incidence and severity of antibody mediated rejection (AMR) analyses
Number of participants with kidney transplant biopsies post baseline | 12 months post baseline, 24 months post baseline
  Number of participants with kidney transplant biopsies post baseline
Proportion of subjects treated for ACR/AMR due to clinical suspicion | 12 months post baseline, 24 months post baseline
  Proportion of subjects treated for ACR/AMR due to clinical suspicion
Number of subjects with de novo anti-donor human leukocyte antigen (HLA) antibodies | 12 months post baseline, 24 months post baseline
  Incidence of de novo anti-donor human leukocyte antigen (HLA) antibodies
First occurrence of graft loss or death post baseline | 12 months post baseline, 24 months post baseline
  First occurrence of graft loss or death at 6, 12 and 24 months post baseline
Number of deaths at 6, 12 and 24 months post baseline | 12 months post baseline, 24 months post baseline
  Incidence of death with graft function at 6, 12 and 24 months post baseline
Incidence of death-censored graft loss post baseline | 12 months post baseline, 24 months post baseline
  Incidence of death-censored graft loss at 12 and 24 months
Compliance with patient-administered subcutaneous abatacept | 12 months post baseline, 24 months post baseline
  Compliance with patient-administered subcutaneous abatacept
Incidence of adverse events | 12 months post baseline, 24 months post baseline
  Incidence of adverse events
Incidence of serious adverse events | 12 months post baseline, 24 months post baseline
  Incidence of serious adverse events
Incidence of events of special interest | 12 months post baseline, 24 months post baseline
  Incidence of events of special interest, including CMV viremia, BKV viremia, and serious infections
Incidence of any malignancy | 12 months post baseline, 24 months post baseline
  Incidence of any malignancy including PTLD
Incidence of subcutaneous injection site complications | 12 months post baseline, 24 months post baseline
  Incidence of subcutaneous injection site complications
Proportion of subjects who develop de-novo, anti-HLA donor specific antibody | 12 months post baseline, 24 months post baseline
  Proportion of subjects who develop de-novo, anti-HLA donor specific antibody

CONTACTS AND LOCATIONS:
Overall Officials: Idelberto R Badell, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital (EUH), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article will be shared, after de identification (text, tables, figures, and appendices) to Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, for individual participant data meta-analysis.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University&amp;amp;amp;amp;#39;s data warehouse but without investigator support other than deposited metadata.
  Individual participant data that underlie the results reported in this article will be shared, after de identification (text, tables, figures, and appendices) to Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, for individual participant data meta-analysis.